CLINICAL TRIAL: NCT02465242
Title: Pupillometry for the Prediction of Neurologic Outcomes in Severe Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Our Lady of the Lake Hospital (Other)
Responsible Party: Principal Investigator, Danielle Tatum, Academic Research Director, Our Lady of the Lake Hospital
Other Study IDs: #8657
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NPi greather than 3: All patients will undergo initial pupillometry evaluation with recording of the NPi in the initial evaluation in the emergency department as per standard evaluation of all trauma patients. If pupils are unequal, group assignment will be determined by lowest pupil reading. Patients with an NPi greater than 3 will be assigned to this group. Pupillometry readings will be gathered for the first 7 days of hospital admission or until discharge. 30, 60, and 90 day post-injury outcomes will be collected.
- NPi less than or equal to 3: All patients will undergo initial pupillometry evaluation with recording of the NPi in the initial evaluation in the emergency department as per standard evaluation of all trauma patients. If pupils are unequal, group assignment will be determined by lowest pupil reading. Patients with an NPi less than or equal to 3 will be assigned to this group. Pupillometry readings will be gathered for the first 7 days of hospital admission or until discharge. 30, 60, and 90 day post-injury outcomes will be collected.

SUMMARY:
Traumatic brain injury (TBI) is a major cause of morbidity and mortality in the US. The CDC states that 1.7 million people sustain a traumatic brain injury each year, with death occurring in 52,000 of these injured patients. It is also estimated that 275,000 yearly require hospitalization. The costs of TBI can be devastating to our society, with the 2010 economic cost estimated to be approximately $76.5 billion. 90% of this cost involves fatal or hospitalized brain injured patients. Furthermore, survivors of traumatic brain injury have high rates of institutionalization, readmission, and disability.

The prediction of prognosis in severe TBI is a difficult problem for physicians. Prognosis evaluation in the acute phase of care varies widely among physicians caring for these patients[3]. With prognosis often in doubt, physicians have difficulty leading families and patients toward the most appropriate treatment which often leads to expensive testing and patient management. The Brain Trauma Foundation has recommended several early indicators of prognosis in severe TBI, including age, hypotension, CT scan features, Glasgow Outcome Scale score, and pupillary diameter with light reflexes. Pupillary diameter and light reflexes have been extensively studied, however accurate measurements of these prognostic factors have not been performed due to a lack of standardized measuring procedure.

A new device has been validated to measure both pupil size and reactivity using infrared pupillometry. This device has also been studied to create the Neurological Pupil Index (NPi) as a measure of pupillary reactivity. The NPi has been shown to correlate with intracranial pressure readings, however there are no studies correlating the pupillometer findings with outcome measures in TBI. This study will prospectively evaluate the pupillometer readings of pupillary size and reactivity (NPi) to test the hypothesis that the NPi is a realiable predictor of 30-day outcomes in patients with severe TBI.

DETAILED DESCRIPTION:
BACKGROUND Pupillary light reflexes have long been used as an important prognostic parameter for predicting outcome following severe TBI. Despite this long history, pupillary assessment remains an inexact science replete with subjectivity and high inter-rater variability. This highlights the need for a reliable, standardized, and accurate measuring procedure.

The NeurOptics NPi-100 Pupillometer is a handheld portable infrared device that allows for objective measurement of pupillary sizes and reflexes. This device utilizes an algorithm derived from multiple measurements taken automatically by the pupillometer to generate the NPi (Neurological Pupil Index). This index allows clinicians to reliably quantify the various aspects of pupillary response to a logical, quantitative scale. Similar devices have demonstrated improvements in both inter- and intra-observer reliability in the assessment of the pupillary response. Although pupillometry has been shown to be a reliable and early indicator of increased intracranial pressure, it is unclear if the results of pupillometry or the NPi can reliably predict functional outcomes in patients with traumatic brain injury.

STUDY OBJECTIVE This is a prospective study designed to determine if the pupillary reflex, as measured by pupillometry and quantified by the NPi, is a reliable prognosticator of both functional outcome and/or mortality in patients with TBI.

STUDY POPULATION The patients to be included in this study will be adults 18 years of age or older who present to the emergency department (ED) with a traumatic brain injury and who are intubated requiring mechanical ventilation.

STUDY PROCEDURES All patients will undergo initial pupillometry evaluation with recording of the NPi in the initial evaluation in the ED as per standard evaluation of all trauma patients. Beyond that, pupillometry and reporting of the NPi will be performed every six (6) hours (Q4) by the bedside nurse throughout the patient's stay in the TNCC. For the long term follow-up phase, functional recovery [as determined by the Functional Independence Measure (FIM) and Functional Assessment Measure (FAM)], Activities of Daily Living (ADL), and Quality of Life (QoL) among the TBI survivors will be assessed when the patients are discharged from the hospital and/or rehabilitation facility. Functional recovery (FIM + FAM) will be assessed at discharge from the TNCC and at 30, 60, and 90 days post-injury. ADL and QoL will be assessed at 90 days post-injury. Vital status will be recorded at discharge from the TNCC and at 90 days post-injury.

POTENTIAL RISK All interventions are usual practice/standard of care within our institution. There is essentially no risk to our patients due to this study.

Because the investigators are maintaining identifiable information for long-term follow-up and assessment, the potential for loss of personal health information exists. To attenuate this risk, all identifiable information will be kept on a password-protected hospital computer in a locked office.

POTENTIAL BENEFIT There is little specific benefit to the individual subjects in this study other than contributing to the advancement of knowledge. A general benefit would be demonstrating the pupillometer to be a reliable predictor of functional outcome of TBI. This would better aid physicians in their prognosis evaluation in the acute phase of care and in deciding the most appropriate treatment for patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older
* Presence of subdural hematoma (SDH), subarachnoid hemorrhage (SAH), epidural hematoma (EDH) or intracerebral hemorrhage (ICH), or cerebral contusion resultant from traumatic brain injury
* Intubated requiring mechanical ventilation

Exclusion Criteria:

* Unable to obtain initial pupillometer reading within six (6) hours of traumatic insult
* History of blindness or enucleation of one or both eyes
* Traumatic injury to one or both eyes such that pupillometry is not possible
* Previous history of known Third Cranial Nerve palsy
* Administration of IV or topical atropine within 6 hours of first pupillometer reading
* Unwilling or unable to consent (or unable to find an appropriate surrogate)
* Pregnant
* History of severe dementia or neurodegenerative disease, mental illnesses requiring long-term institutionalization, severe neuromuscular disorders (Parkinson's disease, Huntington's disease), previous structural brain defect either congenital or due to previous trauma or medical disease, previous anoxic brain injury
* Expected death within 24 hours of enrollment, or desire by patient of family to pursue palliative rather than aggressive, supportive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult trauma patients age 18 years or older with evidence of traumatic brain injury and intubated requiring mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure + Functional Assessment Measure (FIM + FAM) | Time of discharge from ICU, which is typically a duration of 2-3 weeks
  The FIM/FAM is a single outcome measure. The FAM is an adjunct to the FIM and is not meant to stand alone as an assessment measure.

SECONDARY OUTCOMES:
Survival | Patients will be followed for duration of hospital stay, typically a duration of 2-3 weeks, but potentially longer in the case of more severe cases
Time to discharge from acute care facility | Patients will be followed for duration of hospital stay, typically a duration of 2-3 weeks, but potentially longer in the case of more severe cases
Time to discharge to home | Patients will be followed for duration of hospital stay, typically a duration of 2-3 weeks, but potentially longer in the case of more severe cases
FIM + FAM at 30, 60, and 90 days post injury | 30, 60, and 90 days post injury
Activities of daily living (ADL) | 90 days post injury
Quality of Life (QoL) | 90 days post-injury

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Tatum, Ph.D., Principal Investigator — Our Lady of the Lake Hospital
Locations (1):
- Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana, United States